CLINICAL TRIAL: NCT01746979
Title: A Randomized, Double-Blind, Phase III Study of the Efficacy and Safety of Gemcitabine in Combination With TH-302 Compared With Gemcitabine in Combination With Placebo in Previously Untreated Subjects With Metastatic or Locally Advanced Unresectable Pancreatic Adenocarcinoma
Brief Title: Clinical Trial Testing TH-302 in Combination With Gemcitabine in Previously Untreated Subjects With Metastatic or Locally Advanced Unresectable Pancreatic Adenocarcinoma
Acronym: MAESTRO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ImmunoGenesis (Industry)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMR 200592-001; 2012-002957-42 (EudraCT Number)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Results first posted 2017-12-02 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2017-10

CONDITIONS: Metastatic or Locally Advanced Unresectable Pancreatic Adenocarcinoma
Keywords: TH-302; Evofosfamide; Pancreatic Cancer; EMR200592-001
MeSH Terms: conditions — Neoplasm Metastasis; Pancreatic Neoplasms | interventions — TH 302; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine plus TH-302 (Active Comparator)
  Interventions: Drug: TH-302; Drug: Gemcitabine
- Gemcitabine plus placebo (Placebo Comparator)
  Interventions: Drug: Gemcitabine; Drug: Placebo (5 percent dextrose - D5W)

INTERVENTIONS:
Drug: TH-302 — TH-302 will be administered at a dose of 340 milligrams per square meter (mg/m^2) as intravenous infusion over 30 minutes on Day 1, 8 and 15 of every 28-day cycle. Doses will be administered until evidence of progressive disease, intolerable toxicity or subject withdrawal.
  Arms: Gemcitabine plus TH-302
Drug: Gemcitabine — Gemcitabine will be administered at a dose of 1000 (mg/m^2) as intravenous infusion over 30 minutes on Day 1, 8 and 15 of every 28-day cycle. Doses will be administered until evidence of progressive disease, intolerable toxicity or subject withdrawal.
Drug: Placebo (5 percent dextrose - D5W) — TH-302 placebo (5 percent dextrose - D5W) will be administered as intravenous infusion over 30 minutes on Day 1, 8 and 15 of every 28-day cycle. Doses will be administered until evidence of progressive disease, intolerable toxicity or subject withdrawal.
  Arms: Gemcitabine plus placebo

SUMMARY:
This Phase 3 trial is a randomized, double-blind, placebo-controlled trial of gemcitabine in combination with TH-302 compared to gemcitabine in combination with placebo in subjects with locally advanced unresectable or metastatic pancreatic adenocarcinoma. Randomized subjects will receive TH-302 plus gemcitabine or gemcitabine plus placebo in 4-week cycles until there is evidence of progressive disease, intolerable toxicity, or the subject discontinues from the trial for other reasons (for example, withdrawal of consent). The primary efficacy endpoint is overall survival (OS) time. The data cut-off for statistical analyses of the primary and secondary endpoints will be reached when 508 events (deaths) will be reported. No planned interim analyses will be conducted. An Independent Safety Monitoring Board (ISMB) will provide periodic evaluations of the unblinded safety data to ensure subject safety and the validity and scientific merit of the study. A total of 660 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Locally advanced unresectable or metastatic pancreatic ductal adenocarcinoma proven by histology or cytology and previously untreated with chemotherapy or systemic therapy other than:

  * Radiosensitizing doses of 5-fluorouracil;
  * Radiosensitizing doses of gemcitabine if relapse occurred at least 6 months after completion of gemcitabine;
  * Neoadjuvant chemotherapy if relapse occurred at least 6 months after surgical resection;
  * Adjuvant chemotherapy if relapse occurred at least 6 months after completion of adjuvant chemotherapy
* Measurable disease (at least one target lesion outside of previous radiation fields) or non-measurable disease by RECIST v.1.1 criteria
* Documentation of disease progression since any prior therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 3 month
* Acceptable liver, renal function and acceptable hematological status
* Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* New York Heart Association (NYHA) Class III or IV congestive heart failure, myocardial infarction within 6 months prior to the date of randomization, unstable arrhythmia or symptomatic peripheral arterial vascular disease
* Symptomatic ischemic heart disease
* Known brain, leptomeningeal or epidural metastases (unless treated and well controlled for at least 3 months)
* Previous malignancy other than pancreatic cancer in the last 5 years, except for adequately treated non-melanoma skin cancer or pre-invasive cancer of the cervix
* Severe chronic obstructive or other pulmonary disease with hypoxemia
* Major surgery, other than diagnostic surgery, less than or equal to 28 days prior to the date of randomization. Subject must have completely recovered from surgery
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Treatment of pancreatic cancer with radiation therapy or surgery less than or equal to 28 days prior to the date of randomization
* Prior therapy with a hypoxic cytotoxin
* Subjects who participated in an investigational drug or device trial less than or equal to 28 days prior to Day 1 of the first cycle
* Known infection with Human Immunodeficiency Virus (HIV), or an active infection with Hepatitis B or Hepatitis C
* Subjects who have exhibited allergic reactions to a structural compound similar to TH-302 or the drug product excipients or to gemcitabine or its excipients
* Other protocol defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 693 (Actual)
Dates: Start 2012-12; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gualberto, MD, PhD, Study Director — EMD Serono Inc., a subsidiary of Merck KGaA, Darmstadt, Germany
Locations (2):
- Please Contact U.S. Medical Information, Rockland, Massachusetts, United States
- Please Contact Merck Communication Center, Darmstadt, Germany

REFERENCES:
- [Derived] Borad MJ, Reddy SG, Bahary N, Uronis HE, Sigal D, Cohn AL, Schelman WR, Stephenson J Jr, Chiorean EG, Rosen PJ, Ulrich B, Dragovich T, Del Prete SA, Rarick M, Eng C, Kroll S, Ryan DP. Randomized Phase II Trial of Gemcitabine Plus TH-302 Versus Gemcitabine in Patients With Advanced Pancreatic Cancer. J Clin Oncol. 2015 May 1;33(13):1475-81. doi: 10.1200/JCO.2014.55.7504. Epub 2014 Dec 15. PMID 25512461

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine Plus TH-302 | Gemcitabine Plus Placebo
Started | 346 | 347
Completed | 0 | 0
Not Completed | 346 | 347

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine Plus TH-302 | Gemcitabine Plus Placebo | Total
Number analyzed (Participants) | 346 | 347 | 693
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9.70) | 63.8 (9.82) | 64.4 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 168 | 323
  Male | 191 | 179 | 370

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as time from randomization to death or last day known to be alive.
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine Plus TH-302 | Gemcitabine Plus Placebo
Number analyzed (Participants) | 346 | 347
months | 8.9 [7.6 to 9.9] | 7.6 [6.7 to 8.3]

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival is defined as the time from randomization to either first observation of progressive disease or occurrence of death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine Plus TH-302 | Gemcitabine Plus Placebo
Number analyzed (Participants) | 346 | 347
months | 5.5 [4.8 to 5.6] | 3.7 [3.6 to 3.8]

ADVERSE EVENTS:
Groups:
- TH-302: TH-302: TH-302 will be administered at a dose of 340 milligrams per square meter (mg/m^2) as intravenous infusion over 30 minutes on Day 1, 8 and 15 of every 28-day cycle. Doses will be administered until evidence of progressive disease, intolerable toxicity or subject withdrawal.
  Gemcitabine: Gemcitabine will be administered at a dose of 1000 (mg/m^2) as intravenous infusion over 30 minutes on Day 1, 8 and 15 of every 28-day cycle. Doses will be administered until evidence of progressive disease, intolerable toxicity or subject withdrawal.
- Placebo: Gemcitabine: Gemcitabine will be administered at a dose of 1000 (mg/m^2) as intravenous infusion over 30 minutes on Day 1, 8 and 15 of every 28-day cycle. Doses will be administered until evidence of progressive disease, intolerable toxicity or subject withdrawal.
  Placebo (5 percent dextrose - D5W): TH-302 placebo (5 percent dextrose - D5W) will be administered as intravenous infusion over 30 minutes on Day 1, 8 and 15 of every 28-day cycle. Doses will be administered until evidence of progressive disease, intolerable toxicity or subject withdrawal.
Arm/Group | TH-302 | Placebo
Serious Adverse Events (participants affected / at risk) | 341/341 | 338/338
Other Adverse Events (participants affected / at risk) | 341/341 | 338/338
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 (N=341) | Placebo (N=338)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (3)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Bacterial prostatitis (Infections and infestations) | 1 (1) | 0 (0)
Biliary sepsis (Infections and infestations) | 3 (3) | 2 (2)
Biliary tract infection (Infections and infestations) | 2 (3) | 0 (0)
Bronchopneumonia (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 4 (5) | 2 (2)
Device related sepsis (Infections and infestations) | 2 (2) | 0 (0)
Diabetic gangrene (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1)
Fungal oesophagitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 1 (1)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 1 (2)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
Meningoencephalitis herpetic (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic abscess (Infections and infestations) | 0 (0) | 1 (1)
Penile infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 9 (11) | 8 (8)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 5 (5) | 5 (5)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Splenic abscess (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 15 (18) | 16 (18)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (7)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 9 (13)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 19 (25)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (3) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 3 (3)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hemianopia (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 1 (2)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Axillary vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 7 (7)
Embolism (Vascular disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 2 (2)
Acute interstitial pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 11 (11)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (8) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 5 (5) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (11)
Duodenal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 4 (4) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 3 (3) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 3 (4) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (4)
Obstruction gastric (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (2)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (13) | 7 (8)
Bile duct obstruction (Hepatobiliary disorders) | 6 (6) | 3 (3)
Bile duct stenosis (Hepatobiliary disorders) | 5 (5) | 5 (5)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (2)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cholangiectasis acquired (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangiolitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 15 (21) | 12 (12)
Cholangitis acute (Hepatobiliary disorders) | 6 (10) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (2) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 4 (4)
Hepatorenal failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Jaundice (Hepatobiliary disorders) | 4 (5) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 6 (6) | 3 (3)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Yellow skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 4 (4)
Chills (General disorders) | 2 (2) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0)
Device occlusion (General disorders) | 0 (0) | 3 (3)
Disease progression (General disorders) | 2 (2) | 4 (4)
Fatigue (General disorders) | 3 (3) | 2 (2)
General physical health deterioration (General disorders) | 14 (15) | 11 (12)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Injection site extravasation (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2)
Multi-organ failure (General disorders) | 1 (2) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 11 (12) | 14 (15)
Stent malfunction (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3) | 3 (3)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Blood glucose fluctuation (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 4 (4)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 2 (2) | 8 (8)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (5)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prescribed overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TH-302 (N=341) | Placebo (N=338)
Anaemia (Blood and lymphatic system disorders) | 108 (254) | 164 (582)
Leukopenia (Blood and lymphatic system disorders) | 29 (47) | 47 (198)
Neutropenia (Blood and lymphatic system disorders) | 94 (248) | 140 (546)
Thrombocytopenia (Blood and lymphatic system disorders) | 61 (151) | 158 (772)
Decreased appetite (Metabolism and nutrition disorders) | 116 (184) | 117 (205)
Dysgeusia (Nervous system disorders) | 33 (39) | 46 (57)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (44) | 44 (55)
Abdominal pain (Gastrointestinal disorders) | 70 (149) | 65 (110)
Abdominal pain upper (Gastrointestinal disorders) | 38 (58) | 44 (66)
Constipation (Gastrointestinal disorders) | 104 (146) | 104 (171)
Diarrhoea (Gastrointestinal disorders) | 89 (181) | 112 (245)
Nausea (Gastrointestinal disorders) | 150 (320) | 168 (354)
Stomatitis (Gastrointestinal disorders) | 53 (78) | 86 (172)
Vomiting (Gastrointestinal disorders) | 109 (233) | 109 (243)
Alopecia (Skin and subcutaneous tissue disorders) | 23 (30) | 68 (81)
Rash (Skin and subcutaneous tissue disorders) | 46 (65) | 63 (104)
Back pain (Musculoskeletal and connective tissue disorders) | 45 (58) | 30 (35)
Asthenia (General disorders) | 71 (165) | 81 (229)
Fatigue (General disorders) | 106 (219) | 98 (234)
Oedema peripheral (General disorders) | 72 (104) | 64 (87)
Pyrexia (General disorders) | 76 (147) | 64 (104)
Neutrophil count decreased (Investigations) | 29 (94) | 52 (301)
Platelet count decreased (Investigations) | 44 (122) | 100 (476)
White blood cell count decreased (Investigations) | 28 (84) | 55 (263)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No